CLINICAL TRIAL: NCT03403231
Title: INcreasing Veteran EngagemeNT to Prevent Diabetes (INVENT) (CDA 13-267)
Brief Title: INcreasing Veteran EngagemeNT to Prevent Diabetes (INVENT)
Acronym: INVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CDX 15-002; CDA 13-267 (Other Grant/Funding Number: HSR&D)
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Results first posted 2021-06-16 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Prediabetes
Keywords: Veterans; Type 2 diabetes mellitus; Prediabetes; Secure Messaging; Health Promotion; Prevention and Control; Motivation
MeSH Terms: conditions — Prediabetic State; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: The investigators will use a factorial design to test the main effects and a limited number of interaction effects of 5 messaging strategies.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (16):
- Arm 1: Stock messages only (Active Comparator): Participants will only receive the stock messages that encourage following recommended behaviors for reducing the risk for developing diabetes.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 2: Urgency frame message strategy (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with the urgency frame message strategy.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 3: Social norm message strategy (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with the social norm messaging strategy.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 4: Urgency frame and social norm strategies (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with both the urgency frame and social norm messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 5: Implementation Intentions and Urgency Frame (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with both the implementation intentions and urgency frame messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 6: Implementation Intentions and Social Norm (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with both the implementation intentions and social norm messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 7: Implementation Intentions, Urgency Frame & Social Norm (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with the implementation intentions, urgency frame, and social norm messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 8: Implementation Intentions (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with the implementation intentions messaging strategy.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 9: Preference Checklists and Urgency Frame (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with both the preference checklists and urgency frame messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 10: Preference Checklists and Social Norms (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with both the preference checklists and social norm messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 11: Preference Checklists, Urgency Frame & Social Norm (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with the preference checklists, urgency frame, and social norm messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 12: Preference Checklists (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with the preference checklists messaging strategy.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 13: Tailored Aspirations and Urgency Frame (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with both the tailored aspirations and urgency frame messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 14: Tailored Aspirations and Social Norm (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with both the tailored aspirations and social norm messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 15: Tailored Aspirations, Urgency Frame & Social Norm (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with the tailored aspirations, urgency frame, and social norm messaging strategies.
  Interventions: Behavioral: INVENT Secure Messaging Intervention
- Arm 16: Tailored Aspirations (Experimental): Participants will receive messages that encourage following recommended behaviors for reducing the risk for developing diabetes integrated with the tailored aspirations messaging strategy.
  Interventions: Behavioral: INVENT Secure Messaging Intervention

INTERVENTIONS:
Behavioral: INVENT Secure Messaging Intervention — We are proposing a 12 week schedule of weekly Secure Messages and monthly mailings for this intervention. Each study arm represents different combinations of messages a participant will receive.

SUMMARY:
This study will evaluate a VA MyHealtheVet Secure Messaging intervention that uses different intervention messaging strategies designed to increase engagement in behaviors to prevent type 2 diabetes.

The investigators will enroll 144 eligible Veterans into a 12-week MyHealtheVet Secure Messaging intervention. Eligible Veterans include those who are currently using MyHealtheVet secure messaging, meet inclusion/exclusion criteria, and have received an HbA1c test within the last 6 months that meets the ADA/CDC classification for prediabetes. Study participants will be surveyed about their engagement in behaviors to prevent TDM2 and mediators of this engagement. After completing a baseline survey, participants will be randomly assigned to receive different novel presentations of information about ways to prevent T2DM through both Secure Messaging and US Mail. The investigators will test the 5 presentations that each: (1) represent an innovative approach from behavioral economics or health psychology with great promise to increase engagement in behaviors to prevent T2DM among patients with prediabetes; and (2) have not been tested in this setting.

DETAILED DESCRIPTION:
There is tremendous national enthusiasm for translating and disseminating efficacious strategies to prevent type 2 diabetes mellitus (T2DM). Yet, little attention has been devoted to how the investigators can better leverage the processes through which patients receive information about prevention of T2DM to better engage them in such prevention. Further, despite efforts to disseminate structured programs, many patients at high risk for developing T2DM may still be unable or unwilling to access them. In these cases, increasing patient engagement in individually directed lifestyle change or pharmacotherapy is critical. Strategies developed in the fields of behavioral economics and health psychology hold significant promise for improving Veteran engagement in each of these approaches. To date, however, these strategies have rarely been translated into real-world settings where they could benefit Veterans. This novel work will address this critical gap and could transform communication with Veterans about prevention in ways that will improve their health outcomes.

The following 5 strategies will be implemented in the weekly messages that study participants will receive: (1) tailoring to aspirations in life; (2) implementation intentions; (3) preference checklists; (4) urgency framing; (5) social norms. The investigators will implement these strategies alone and in combination in a 16-arm factorial design experiment.

ELIGIBILITY:
Inclusion Criteria:

1. HbA1c test within the past 6 months that meets the ADA/CDC requirements for prediabetes.
2. Currently registered in the VA's MyHealtheVet Secure Messaging System
3. Receiving care within the Ann Arbor VA Healthcare System

Exclusion Criteria:

1. Completed more than 4 VA MOVE! classes in the last year (or other evidence of another recent weight loss program)
2. Are trying to lose weight and are very physically active
3. Are >75 years of age
4. Are pregnant or plan to be
5. Are taking Metformin
6. Have participated in the FINDIT study (this study's predecessor under the same grant funding)
7. Have been hospitalized or received rehab for stroke or myocardial infarction within past 6 months
8. Have received chemotherapy for cancer in the past 6 months
9. Self-report or have any International Classification of Diseases (ICD-9/10) codes for:

   * Diabetes
   * Dementia
   * Major functional limitations
   * Cirrhosis
   * Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage 4 chronic obstructive pulmonary disease (COPD)
   * End stage renal disease (ESRD)
   * New York Heart Association (NYHA) class III or IV congestive heart failure (CHF)

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey T. Kullgren, MD MPH MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans that met preliminary study eligibility criteria were mailed a letter about the study and were contacted by a Research Assistant 7-10 days later by phone to gauge their participation interest.
Pre-assignment Details: The population consisted of prediabetic Veterans ages 75 and younger, had access to VA MyHealtheVet Secure Messaging, and met inclusion and exclusion criteria. Those that did not complete the Baseline Survey or did not have consistent internet access to use MyHealtheVet Secure Messaging were not randomized and thus excluded from analysis.
Period: Overall Study
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Started | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled study participants with a diagnosis of prediabetes that were randomized to 1 of 16 study arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 3 | 4 | 7 | 3 | 6 | 7 | 6 | 4 | 6 | 3 | 4 | 4 | 7 | 3 | 74
  >=65 years | 4 | 7 | 6 | 5 | 2 | 6 | 3 | 2 | 3 | 5 | 3 | 6 | 5 | 5 | 2 | 6 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (13.4) | 66 (8.3) | 62.1 (13.1) | 62.1 (8.9) | 55.6 (10.2) | 64.2 (9.0) | 63.3 (5.8) | 57.4 (10.9) | 62.4 (5.5) | 60.1 (10.3) | 62.1 (6.4) | 64.7 (9.0) | 63.1 (9.9) | 61.2 (10.0) | 57.1 (7.6) | 61.6 (11.3) | 61.3 (9.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 9 | 8 | 8 | 8 | 7 | 8 | 7 | 8 | 8 | 6 | 6 | 9 | 9 | 9 | 9 | 7 | 126
  Female | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 3 | 3 | 0 | 0 | 0 | 0 | 2 | 17
  Transgender | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 9 | 9 | 8 | 7 | 9 | 9 | 9 | 9 | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 9 | 139
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 9
  White | 8 | 8 | 8 | 7 | 7 | 8 | 8 | 6 | 8 | 8 | 8 | 7 | 7 | 6 | 8 | 8 | 120
  More than one race | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 144

OUTCOME MEASURES:

1. Primary Outcome: Engagement in Recommended Behaviors to Prevent Type 2 Diabetes
Description: The investigators will use survey and medical record data to evaluate changes in participants' engagement in recommended behaviors to prevent type 2 diabetes.
Time Frame: 3 months
Population: The population consisted of prediabetic Veterans ages 75 and younger, had access to VA MyHealtheVet Secure Messaging, and met inclusion and exclusion criteria at the time of enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Participants
  Engaged in recommended behaviors | 2 | 5 | 5 | 2 | 2 | 3 | 2 | 2 | 6 | 4 | 2 | 4 | 2 | 2 | 4 | 0
  Did not engage in recommended behaviors | 6 | 4 | 4 | 7 | 6 | 5 | 7 | 5 | 3 | 5 | 7 | 5 | 5 | 6 | 5 | 7
  Unknown | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2

2. Secondary Outcome: Motivation to Prevent Type 2 Diabetes
Description: The investigators will use survey data to evaluate mean change in motivation level to prevent diabetes between baseline and 3-months. The Treatment Self-Regulation Questionnaire (TSRQ) was included in the survey and respondents were asked about their level of motivation from 1 (Not at all motivated) to 10 (Highly motivated).
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Score on a scale | .375 (2.326) | -1.222 (2.438) | -0.444 (1.333) | -0.222 (1.394) | 0.429 (2.225) | 0.000 (0.7071) | 0.333 (1.500) | -1.143 (2.673) | -2.000 (3.122) | -0.666 (1.323) | -0.333 (2.540) | -0.222 (1.986) | -1.166 (1.472) | -0.286 (0.9512) | -0.555 (1.333) | 0.857 (2.116)

3. Secondary Outcome: Importance of Preventing Type 2 Diabetes
Description: The investigators will use survey data to evaluate mean changes in level of importance of preventing diabetes from baseline to 3 months. The Treatment Self-Regulation Questionnaire (TSRQ) was included in the survey and respondents were asked about their level of perceived importance from 1 (Not at all important) to 10 (Extremely important).
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Score on a scale | -0.625 (1.847) | -0.889 (2.028) | -0.444 (1.740) | -0.222 (1.563) | 0.714 (2.430) | 0.000 (0.500) | -0.500 (2.000) | -1.571 (2.070) | -1.111 (2.934) | -0.333 (1.118) | -0.667 (2.000) | 0.667 (1.936) | -0.333 (2.582) | 0.429 (0.976) | -2.333 (2.236) | 0.286 (1.254)

4. Secondary Outcome: Use of Medication for T2DM Prevention
Description: The investigators will use medical record data and survey data to evaluate whether participants began the use of medication for T2DM prevention from baseline to 3 months.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Participants
  Taking medication | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Not taking medication | 7 | 8 | 8 | 9 | 8 | 8 | 9 | 7 | 9 | 9 | 8 | 9 | 7 | 8 | 8 | 7
  Unknown | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2

5. Secondary Outcome: Perception for Risk for T2DM
Description: The investigators will use survey data to evaluate mean changes in perception of risk for T2DM from baseline to 3 months. The Adriaanse T2DM Risk Perception Scale, which was included in the survey, measured self-assessed risk perception from 0 denoting no choice of developing T2DM to 100 denoting absolute confidence in developing T2DM
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Score on a scale | -8.750 (8.345) | -1.111 (13.642) | 6.667 (15.000) | -4.444 (13.333) | 0.000 (17.321) | 1.111 (9.280) | -5.556 (40.035) | 10.000 (20.000) | 7.778 (24.889) | -3.333 (11.180) | 8.333 (24.238) | -2.222 (28.626) | 5.000 (25.100) | 10.000 (21.602) | 3.333 (33.166) | 10.000 (25.166)

6. Secondary Outcome: Knowledge of Strategies to Prevent T2DM
Description: The investigators will use survey data to evaluate changes in knowledge of strategies to prevent Type 2 Diabetes between baseline and 3-month assessment. Respondents were given 3 open-ended questions to report things they could do to prevent diabetes. Each respective response to the 3 questions were coded and scored according to whether they indicated engagement in the following activities: weight loss, physical activity, use of metformin, or enrollment into a diabetes prevention program. Each question denoted with a positive response were coded with 1 whereas those that did not were coded as a 0. The three questions were summed into a final score ranging from 0 (no report of engagement in the aforementioned healthy activities) with the worst outcome to 3 (a report of 3 of the 4 aforementioned healthy activities) with the best outcome. The final scores were generated based on the mean difference between baseline and 3-month scores.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Score on a scale | 0 (1.069) | -0.222 (0.667) | -0.222 (0.833) | -0.222 (0.972) | 0.125 (0.641) | -0.444 (0.882) | 0.444 (0.726) | 0.429 (0.535) | 0.333 (0.866) | 0.333 (0.707) | 0.889 (0.928) | -0.333 (0.500) | 0.143 (0.378) | 0 (0.535) | 0.778 (0.833) | 0.286 (0.488)

7. Secondary Outcome: Participation in Weight-related Wellness Programs
Description: The investigators will use survey data to evaluate how many participants enrolled in weight-related wellness programs from baseline to 3 months.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Participants
  Participation in weight-related wellness programs | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  No participation in weight-related wellness programs | 8 | 9 | 9 | 9 | 7 | 8 | 9 | 7 | 9 | 9 | 9 | 8 | 7 | 8 | 8 | 7
  Unknown | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2

8. Secondary Outcome: Weight Loss Behaviors
Description: The investigators will use survey data to evaluate changes in weight loss behaviors at the 3-month post intervention assessment.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Participants
  Losing weight | 2 | 5 | 5 | 2 | 3 | 4 | 2 | 3 | 4 | 4 | 2 | 5 | 1 | 4 | 1 | 0
  Gaining weight | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Stable and satisfied | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Stable and lose | 5 | 2 | 4 | 6 | 4 | 3 | 5 | 3 | 3 | 5 | 7 | 3 | 5 | 3 | 6 | 6
  Stable and gain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Unknown | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2

9. Secondary Outcome: Physical Activity
Description: The investigators will use survey data to evaluate changes in physical activity after the 3-month post intervention assessment. The International Physical Activity Questionnaire - Short Form (IPAQ-SF) was used to measure physical activity change. Respondents were asked to report how many hours and minutes within the past week they completed of vigorous physical activity, moderate physical activity, and brisk walking. The total sum of minutes for these three questions were subsequently coded into a yes/no binary variable for whether respondents met a recommended 150 minutes of overall physical activity within 7 days of being assessed. The values provided reflect a proportion of respondents that met or exceeded the 150 minute threshold of overall physical activity based on the newly generated variable that combined total minutes of vigorous physical activity, moderate physical activity, and brisk walking.
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9
Participants
  150 minutes or more physical activity per week | 5 | 4 | 6 | 7 | 4 | 5 | 6 | 6 | 6 | 7 | 6 | 8 | 3 | 6 | 4 | 2
  Less than 150 minutes or more of physical activity per week | 4 | 5 | 3 | 2 | 5 | 4 | 3 | 3 | 3 | 2 | 3 | 1 | 6 | 3 | 5 | 7

ADVERSE EVENTS:
Time Frame: 3-months
Description: Adverse events information was collected from participants if they reported events during phone correspondence with a Research Assistant related to the brief intervention or 3-month assessment.
Arm/Group | Arm 1: Stock Messages Only | Arm 2: Urgency Frame Message Strategy | Arm 3: Social Norm Message Strategy | Arm 4: Urgency Frame and Social Norm Strategies | Arm 5: Implementation Intentions and Urgency Frame | Arm 6: Implementation Intentions and Social Norm | Arm 7: Implementation Intentions, Urgency Frame & Social Norm | Arm 8: Implementation Intentions | Arm 9: Preference Checklists and Urgency Frame | Arm 10: Preference Checklists and Social Norms | Arm 11: Preference Checklists, Urgency Frame & Social Norm | Arm 12: Preference Checklists | Arm 13: Tailored Aspirations and Urgency Frame | Arm 14: Tailored Aspirations and Social Norm | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm | Arm 16: Tailored Aspirations
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 0/9 | 1/9 | 0/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: Stock Messages Only (N=9) | Arm 2: Urgency Frame Message Strategy (N=9) | Arm 3: Social Norm Message Strategy (N=9) | Arm 4: Urgency Frame and Social Norm Strategies (N=9) | Arm 5: Implementation Intentions and Urgency Frame (N=9) | Arm 6: Implementation Intentions and Social Norm (N=9) | Arm 7: Implementation Intentions, Urgency Frame & Social Norm (N=9) | Arm 8: Implementation Intentions (N=9) | Arm 9: Preference Checklists and Urgency Frame (N=9) | Arm 10: Preference Checklists and Social Norms (N=9) | Arm 11: Preference Checklists, Urgency Frame & Social Norm (N=9) | Arm 12: Preference Checklists (N=9) | Arm 13: Tailored Aspirations and Urgency Frame (N=9) | Arm 14: Tailored Aspirations and Social Norm (N=9) | Arm 15: Tailored Aspirations, Urgency Frame & Social Norm (N=9) | Arm 16: Tailored Aspirations (N=9)
Diagnosis of Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-03-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03403231/Prot_000.pdf